CLINICAL TRIAL: NCT04211194
Title: The Orange County Bleeding Consortium (OCBC): Registry of Patients Undergoing Endoscopic Procedures for Upper Gastrointestinal Bleeding in AdventHealth Hospitals in Central Florida
Brief Title: Registry for Upper Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1494617
Record Dates: First submitted 2019-10-30; First posted 2019-12-26 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Peptic Ulcer Hemorrhage; Peptic Ulcer, Acute With Hemorrhage
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Peptic Ulcer | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with upper gastrointestinal bleeding: Patients with upper gastrointestinal bleeding undergoing endoscopic procedures at AdventHealth Hospitals in Central Florida
  Interventions: Procedure: Upper GI Endoscopy

INTERVENTIONS:
Procedure: Upper GI Endoscopy — Patients with upper gastrointestinal bleeding undergoing endoscopic therapy. Information regarding the need for interventional radiology procedures or surgical interventions will also be collected in patients in whom endoscopic therapy is not successful.

SUMMARY:
This project aims to evaluate the data on all patients undergoing endoscopic therapy for upper gastrointestinal bleeding.

DETAILED DESCRIPTION:
This project is being performed to evaluate the outcomes of patients undergoing endoscopic procedures for upper gastrointestinal bleeding at all AdventHealth hospitals in Central Florida. This information will enable quality control of patients undergoing treatment for upper gastrointestinal bleeding across all campuses in the AdventHealth system in Central Florida and hence improve the delivery ot care extended to the investigator's patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or greater
* Patient is undergoing endoscopic treatment for upper gastrointestinal bleeding

Exclusion Criteria:

* Under the age of 18
* Patient not undergoing endoscopic treatment for upper gastrointestinal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will come from patient who are undergoing endoscopic treatment for upper gastrointestinal bleeding at AdventHealth Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 2999 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Mortality Rate | 30 days
  Mortality rate from upper gastrointestinal bleeding and from any etiology

SECONDARY OUTCOMES:
Rate of Reintervention | 30 days
  Need for repeat endoscopic treatment for upper gastrointestinal bleeding
Rate of Recurrence | 30 days
  Recurrence of upper gastrointestinal bleeding following endoscopic treatment
Rate of Readmission | 30 days
  Need for readmission to hospital for treatment of upper gastrointestinal bleeding
Length of hospital stay | 30 days
  Length of hospitalization from index endoscopic procedure to discharge
Costs | 30 days
  Total hospital costs from admission for upper gastrointestinal bleeding
Treatment success | 30 days
  Successful treatment of upper gastrointestinal bleeding using endoscopic therapy as determined by a yes/no answer.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth Orlando
Locations (1):
- Center for Interventional Endoscopy, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No